CLINICAL TRIAL: NCT06678295
Title: Contributions of Self-Focused Attention to Early Warning Indicators of Cognitive Behavioral Therapy Non-Response
Brief Title: Individual Factors of CBT Underlying Success
Acronym: I-FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Angela Fang, Associate Professor of Psychology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019785; R01MH133581 (NIH)
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Social Anxiety Disorder; Body Dysmorphic Disorder
Keywords: Body Dysmorphic Disorder; Social Anxiety Disorder; Social Phobia; Self focused attention; fMRI; CBT; Cognitive Behavior Therapy; BDD; SAD; Neuroimaging
MeSH Terms: conditions — Phobia, Social; Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive behavioral therapy (Experimental): Twelve weekly sessions of individual cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Twelve weekly sessions of individual cognitive behavioral therapy

SUMMARY:
The purpose of this study is to understand why some individuals respond fully to cognitive behavioral therapy and others do not, based on multiple sources of data such as neural, neurocognitive, clinical, and self-report data.

DETAILED DESCRIPTION:
The investigators are conducting this research to evaluate the reliability and construct validity of measures of self-focused attention (SFA) across neural, neurocognitive, and self-report levels of analysis as well as examine whether early changes in the SFA biomarker are associated with CBT non-response.

This will be looked at in a clinical population consisting of individuals with social anxiety disorder (SAD) and body dysmorphic disorder (BDD) compared to healthy volunteers. This study employs an open clinical trial for cognitive behavioral therapy with pre-, mid- and post-treatment neuroimaging scans, clinical interviews, neurocognitive, behavioral, and self-report assessments. Clinical participants will be invovled for 3.5 months and complete 12 CBT sessions and 4 fMRI scans. Control participants will not participate in CBT treatment and will complete 3 fMRI scans across a 3.5 month period. About 160 people will take part in this research study, all at the University of Washington (UW). This will include 110 clinical participants and 50 healthy control participants.

ELIGIBILITY:
Inclusion Criteria:

Clinical sample (N=110):

1. Men and women, age 18-45
2. Treatment-seeking individuals who meet criteria for a primary DSM-5 diagnosis of primary social anxiety disorder (SAD) or body dysmorphic disorder (BDD) based on the SCID-5-RV
3. Fluent in English and willing to provide informed consent.

Control sample (N=50):

1. Men and women, age 18-45
2. No current or lifetime history of psychiatric disorders, as assessed using the SCID-5-RV
3. Meet criteria for low levels of anxiety (GAD-7 score of <8) and depression (PHQ-9 score <10)
4. Fluent in English and willing to provide informed consent

Exclusion Criteria:

All groups:

1. Score < 80 based on WRAT5 Word Reading Subtest
2. fMRI contraindications (e.g., electronic medical devices such as pacemakers, implanted defibrillators, etc.; metal implants not approved for MRI; pregnancy; claustrophobia)

2. Active suicidal or homicidal ideation, or any features requiring a higher level of care 3. Lifetime history of manic or hypomanic episode, psychotic symptoms, traumatic brain injury, neurological disorder, pervasive developmental disorder, or attention deficit-hyperactivity disorder; active alcohol or substance use disorder in the past 6 months 4. Current use of psychotropic medications, except antidepressants taken at a stable dose for 3 months prior to study baseline 5. Previous CBT non-responder or current CBT

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Trait SFA assessed by the Public Self-Consciousness Scale- Revised (SCS-R) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  Participants will complete the 7-item self-report Public SCS-R measure to assess trait self-focused attention.
Functional connectivity between the Default Mode and Dorsal Attention Networks (DMN-DAN) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 6, Post-treatment
  Participants will complete an MRI scan comprising both task and resting state fMRI to derive a measure of intrinsic functional connectivity between DMN and DAN using general functional connectivity.
Anxiety symptom severity, assessed by the Structured Interview Guide for Hamilton Anxiety Scale (SIGH-A) and the Generalized Anxiety Disorder (GAD-7) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  The SIGH-A is a 14-item clinician-rated assessment of past-week anxiety symptom severity. Scores on the SIGH-A (together with scores on the CGI-I) will be used to calculate a categorical measure of treatment response (e.g., Remitters, Partial Responders, or NonResponders). SIGH-A items will be adapted to accommodate anxiety symptoms in a transdiagnostic sample (e.g., accounting for specific disorder-relevant fears in item 3, such as fear of negative appearance evaluation in BDD). Generalized Anxiety Disorder (GAD-7) is a 7-item self-report measure of severe anxiety
Anxiety symptom severity, assessed by the Generalized Anxiety Disorder (GAD-7) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  Generalized Anxiety Disorder (GAD-7) is a 7-item self-report measure of severe anxiety
Symptom severity associated with primary disorder, assessed by self-report versions of the Liebowitz Social Anxiety Scale (LSAS SR). | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment. DSM5 Cross Cutting: Baseline (T-2weeks), Repeat Baseline (T0), Post-treatment
  Total scores from the LSAS-SR will be used toward calculating a categorical measure of treatment response (e.g., Remitters, Partial Responders, or NonResponders). Scores will also be examined as a dimensional measure of symptom severity change during treatment based on the participant's primary disorder. Standardized change scores will be calculated based on the pretreatment score on the selected measure.
Symptom severity associated with primary disorder, assessed by self-report version of the Yale-Brown Obsessive-Compulsive Scale Modified for BDD (BDD-YBOCS SR). | Across the span of 3 1/2 months: BDD-YBOCS: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment. DSM5 Cross Cutting: Baseline (T-2weeks), Repeat Baseline (T0), Post-treatment
  Total scores from the BDD-YBOCS-SR will be used toward calculating a categorical measure of treatment response (e.g., Remitters, Partial Responders, or NonResponders). Scores will also be examined as a dimensional measure of symptom severity change during treatment based on the participant's primary disorder. Standardized change scores will be calculated based on the pretreatment score on the selected measure.
DSM5 Cross Cutting Form | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment. DSM5 Cross Cutting: Baseline (T-2weeks), Repeat Baseline (T0), Post-treatment
  The DSM-5 Cross Cutting Measure is a 24-item self-report measure that assesses symptom related problems over the past 2 weeks.

SECONDARY OUTCOMES:
Trait rumination assessed by the Ruminative Responses Scale (RRS) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 6, Post-treatment
  Participants will complete the 22-item self-report RRS measure to assess trait levels of rumination.
Trait worry assessed by the Penn State Worry Questionnaire (PSWQ) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 6, Post-treatment
  Participants will complete the 16-item self-report PSWQ measure to assess trait worry.
Reaction times during Self trials in Self-Other Task | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 6, Post-treatment
  Participants will complete the Self-Other fMRI task and reaction time responses assessed simultaneously during fMRI will be examined as a measure of self-referential processing.
Alerting, orienting, and attentional control reaction time scores on the Attention Network Test (ANT) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  Participants will complete the Attention Network Test, which is a well-validated neurocognitive assay of general attentional mechanisms (alerting, orienting, and attentional control).
Depression severity, as assessed by the Quick Inventory of Depressive Symptomatology (QIDS-SR) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  The QIDS SR is a 16-item self-report measure of depressive symptom severity.
Depression severity, as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Across the span of 3 1/2 months: PHQ-9: Baseline (T-2weeks), Repeat Baseline (T0), and Weekly starting from Week 1.
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item, self-report measure of depression
Insight, as assessed by the Brown Assessment of Beliefs Scale (BABS) | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 3, Week 6, Week 9, Post-treatment
  The BABS is a 7-item clinician-rated instrument of insight and delusionality designed to assess delusions across a wide range of disorders.
Disability, assessed by the Sheehan Disability Scale (SDS). | Across the span of 3 1/2 months: Baseline (T-2weeks), Repeat Baseline (T0), Week 6, Post-treatment.
  The SDS is a 5-item self-report measure of disability in work/school, social life, and family life.
Disability, assessed by the World Health Organization Disability Assessment Schedule (WHODAS) | Across the span of 3 1/2 months: Baseline (T-2 weeks), Repeat Baseline (T0), Post-treatment
  The WHODAS is a 12-item self-report measure of health-related difficulties
Homework compliance, assessed by a modified version of the Patient Exposure/Response Prevention Adherence Scale (PEAS) | Weekly starting from Week 1 to Week 12
  The Modified PEAS is a therapist-rated measure of homework compliance for exposure and nonexposure-related homework
Credibility and expectancies for treatment, assessed by the Credibility and Expectancies Questionnaire (CEQ) | Week 3
  The CEQ is a 6-item self-report measure of patient's beliefs about the credibility of treatment and expectancies for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fang, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No